CLINICAL TRIAL: NCT01195922
Title: A Pilot Trial Targeting mTOR as a Novel Mechanism-Based Neoadjuvant Therapy for Head and Neck Cancer
Brief Title: Rapamycin Therapy in Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100180; 10-D-0180 (Other: NIHCC)
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Results first posted 2017-01-19 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-10

CONDITIONS: Mouth Neoplasms; Head and Neck Neoplasms; Tongue Neoplasms; Carcinoma, Squamous Cell
Keywords: Head and Neck Squamous Cell Carcinoma; Oral Cancer; mTOR Inhibitors; Targeted Therapies; Signal Transduction Inhibitors; Head and Neck Cancer; Squamous Cell Carcinoma; Tongue Cancer
MeSH Terms: conditions — Mouth Neoplasms; Head and Neck Neoplasms; Tongue Neoplasms; Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sirolimus (Experimental): Subjects will be treated with sirolimus 21 days
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — 21 evaluable subjects will take rapamycin (sirolimus) orally once per day for 21 days. Before and after dosing tumor assessments to include: photographs, CT & amp; PET scans will be done for tumor measurement.
  Other Names: Rapamycin

SUMMARY:
Background:

- Advanced-stage head and neck cancer (head and neck squamous cell carcinoma [HNSCC]) has moderately successful treatment outcomes, usually involving surgery as part of the standard treatment. Researchers are investigating the use of the drug rapamycin to prevent tumor growth in HNSCC, and are interested in using it to treat individuals with HNSCC that has not been treated previously with other drugs, radiation, or surgery.

Objectives:

- To evaluate the usefulness of rapamycin in decreasing tumor size prior to surgery for head and neck squamous cell carcinoma.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with advanced head and neck squamous cell carcinoma that has not yet been treated.

Design:

* Participants will be screened with a physical examination, medical history, blood tests, and imaging studies.
* Approximately 1 month before scheduled surgery, participants will begin to receive rapamycin. Participants will take rapamycin once daily for 21 days, followed by a 7-day period without the drug.
* During the 21-day rapamycin treatment, participants will have weekly study visits to provide blood and urine samples and have possible tumor biopsies and imaging studies such as x-rays or tumor photographs. Participants will have additional study visits for tests 1 day and 1 week after the end of rapamycin treatment, followed by HNSCC surgery.
* Participants will have a final visit to provide blood samples 30 days after surgery.
* Participants medical records will be reviewed 1 year after surgery; however, participants will not need to have further study visits at this time.

DETAILED DESCRIPTION:
BACKGROUND:

* The five-year survival rate for head and neck squamous cell carcinoma (HNSCC) has remained at approximately 50% for more than three decades.
* In HNSCC, the AKT-mTOR-pS6 pathway is aberrantly activated and promotes tumorigenesis and metastasis.
* Rapamycin is the most extensively studied mTOR inhibitor for which therapeutic daily oral dose and schedule, pharmacologic levels in blood, and safety have been established.
* Inhibition of mTOR by rapamycin causes the rapid apoptotic death of HNSCC tumor xenografts and decreases the tumor burden and prolongs the survival of mice harboring early and advanced oral and skin SCC lesions in a variety of experimental cancer models.
* Preliminary evidence suggests that mTOR inhibitors cause tumor shrinkage and improved tumor margins in HNSCC patients.

OBJECTIVES:

* The primary objectives are to evaluate the following for patients with HNSCC given rapamycin as neoadjuvant treatment prior to surgery or chemoradiation:

  * Whether therapeutic activities of rapamycin lead to inhibition of mTOR complexes, mTORC1 and mTORC2, as assessed by the change in levels of pS6 and pAkt473 measured by immunohistochemistry (IHC) in tumor samples and by Western blotting in peripheral blood mononuclear cells (PBMCs) and reduce tumor cell proliferation, as judged by IHC for Ki-67 in tumor samples.
  * Antitumor activity in terms of objective response.
* Secondary objectives include safety evaluation of rapamycin therapy, exploratory studies of possible effects of rapamycin on tumor size, dynamic CT perfusion, and FDG-PET; and evaluation of tumor proliferation, apoptosis, microvessel density, and molecular changes associated with these effects. Survival status, recurrence of disease, metastases, and adverse events/serious adverse events, including complications of wound healing, which are related to rapamycin therapy will also be assessed for 360 days after surgery or chemoradiation through medical record review.

ELIGIBILITY:

* Males and females age 18 years and older
* Previously untreated HNSCC of the oral cavity or oropharynx
* Clinical stage II, III, or IVA disease without distant metastasis
* Definitive therapy to include surgical resection or chemoradiation for curative purposes
* Life expectancy greater than six months

STUDY DESIGN:

* Pilot, single arm, open-label, interventional neoadjuvant clinical trial.
* Twenty one evaluable subjects will take rapamycin (sirolimus) orally once per day for 21 days.
* Before and after dosing, the tumor will be photographed and biopsied, peripheral blood mononuclear cells (PBMCs) will be collected, and computed tomography and positron emission tomography scans will be performed.
* Surgical or chemoradiation treatment, which is being provided outside of this protocol, will be conducted after Day 28 and when rapamycin levels are less than or equal to 3 nanograms per milliter.
* Subjects will be followed by medical record review for 360 days after surgery or chemoradiation to assess 1) survival, 2) recurrence of disease, 3) metastases, and 4) adverse events/serious adverse events that are related to rapamycin therapy, including complications of wound healing and infections due to immune compromise.
* Levels of pS6 and pAkt473 in tumor tissue and PBMCs and Ki-67 in tumor tissue before and after rapamycin therapy will be determined by immunohistochemistry and by Western blotting. Computed tomography (CT) and positron emission tomography (PET) scans of the head, neck, and chest region with and without contrast will be performed within 7 days prior to the first rapamycin administration. One day after the last administration of rapamycin the CT and PET scans (head and neck region only) with contrast will be repeated.
* A single stage design will be used based on response defined as > 25% tumor shrinkage. A Wilcoxon signed rank test will be used to compare levels of pS6, pAkt473, and Ki-67 before and after rapamycin therapy. As part of secondary analysis, the number of subjects achieving a best response of complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 will also be summarized.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Males and females and members of any race or ethnic group who meet the eligibility criteria may participate in this trial.

INCLUSION CRITERIA:

Participants must meet all of the following inclusion criteria:

1. Age 18 years and older
2. Histologically confirmed previously untreated squamous cell carcinoma o f the oral cavity or oropharynx accessible for biopsy
3. Clinical stage II, III, or IVA disease without distant metastasis, as defined by the American Joint Committee on Cancer Staging System, Seventh edition.
4. Definitive therapy to include surgical resection or chemoradiation for curative purposes
5. Life expectancy o f greater than 6 months
6. Eastern Cooperative Oncology Group ( ECOG) performance status of 0 or 1
7. Willing and able to provide written informed consent

EXCLUSION CRITERIA:

Participants who meet any of the following criteria are not eligible for enrollment:

1. Surgical resection or chemoradiation of the HNSCC is contraindicated
2. Prior head or neck squamous cell carcinoma within 5 years, except for previously treated skin cancer
3. Received chemotherapy targeted monoclonal antibody therapy or investigational therapy within 30 days prior to enrollment
4. Previous radiation therapy to the head or neck
5. No measurable tumor remaining after prior biopsy or negative margins from prior biopsy
6. Inadequate hematologic, renal or liver function within l4 days prior to the first rapamycin dosing visit, as defined by:

   1. Absolute neutrophil count less than 1.5 times 10 (9)/L
   2. CD4 count < 400 (to account for natural fluctuations in CD4 levels, participants with at least one CD4 count (Bullet) 400 within 14 days prior to dosing will not be excluded)
   3. Platelet count less than 100 times 10(9)/L
   4. Hemoglobin less than l0 g/dL (eligibility level for hemoglobin may be reached by transfusion)
   5. AST, ALT or bilirubin greater than 1.5 times the upper limit of local lab normal values
   6. Total cholesterol level greater than 350 mg/dL
   7. Triglyceride level greater than 400 mg/dL
   8. International Normalized Ratio (INR) greater than 1.5
   9. Serum creatinine greater than 1.5mg/dL
7. Active hepatitis or HBV or HCV infection
8. Women who are pregnant or lactating (female of child-bearing age must be abstinent or use a barrier type birth control method throughout the study)
9. Presence of any contraindications to rapamycin therapy, including HlV-protease inhibitors and drugs or agents that are modulators of cytochrome P-450 3A4 (CYP3A4) and p-glycoprotein(P-gp)
10. Hypersensitivity to rapamycin

11 .Has received live vaccine (such as influenza nasal vaccine measles mumps, rubella, oral polio, B CG, yellow fever, varicella, or TY2la typhoid) in the past 30 days or has plans to take a live vaccine in the next 3 months

12. Any cognitive impairment that limits the subject s or the subject s legally authorized representative s ability to understand the protocol, provide informed consent or assent, or to comply with the protocol procedures

13.Unable or unwilling to comply with the requirements of the protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-08; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janice S Lee, DDS, MD, Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Murray T, Thun MJ. Cancer statistics, 2008. CA Cancer J Clin. 2008 Mar-Apr;58(2):71-96. doi: 10.3322/CA.2007.0010. Epub 2008 Feb 20. PMID 18287387
- [Background] Forastiere A, Koch W, Trotti A, Sidransky D. Head and neck cancer. N Engl J Med. 2001 Dec 27;345(26):1890-900. doi: 10.1056/NEJMra001375. No abstract available. PMID 11756581
- [Background] Agulnik M, da Cunha Santos G, Hedley D, Nicklee T, Dos Reis PP, Ho J, Pond GR, Chen H, Chen S, Shyr Y, Winquist E, Soulieres D, Chen EX, Squire JA, Marrano P, Kamel-Reid S, Dancey J, Siu LL, Tsao MS. Predictive and pharmacodynamic biomarker studies in tumor and skin tissue samples of patients with recurrent or metastatic squamous cell carcinoma of the head and neck treated with erlotinib. J Clin Oncol. 2007 Jun 1;25(16):2184-90. doi: 10.1200/JCO.2006.07.6554. PMID 17538163
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-D-0180.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the National Institute of Health (NIH) as well as the Medical University of South Carolina (MUSC). Recruitment began 5/16/2011 with a total of 37 subjects consented; 34 at MUSC and 3 and NIH. Of the 37 consented, 16 subjects received study intervention and completed the study.
Pre-assignment Details: 37 participants signed consent, 16 participants received study drug.
Groups:
- Sirolimus: Rapamycin (sirolimus), dispensed as either tablets or an oral solution for patients with dysphagia was administered orally as a single loading dose of 15 mg on the first day and 5 mg once a day for the next 20 days. Dose reductions to 3 mg by mouth once per day were implemented if levels of rapamycin > 20 ng/ml occurred on Days 8 or 15.
Period: Overall Study
Arm/Group | Sirolimus
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Sirolimus: Rapamycin (sirolimus), which will be dispensed as either tablets or an oral solution for patients with dysphagia (see Section 0), will be administered orally as a single loading dose of 15 mg on the first day and 5 mg once a day for the next 20 days. Serum rapamycin levels will be obtained on Days 8, 15, 22, and 28 (if rapamycin is > 3 ng/ml at Day 28, the subject will return daily, or as is convenient, for testing until rapamycin is ≤ 3 ng/ml). Dose reduction to 3 mg by mouth once per day will occur if trough levels of rapamycin > 20 ng/ml occur on Days 8 or 15 (see Appendix A, Study Calendar for visit windows). If a dose is decreased at Day 8, it will not be increased at Day 15 regardless of serum rapamycin levels. If subjects receiving 3 mg have levels > 20 ng/ml at Day 15, rapamycin will be reduced to 2 mg once per day. Rapamycin will cease on Day 21 regardless of level.
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
Age, Continuous [Median (Standard Deviation); unit: years] | 63 (11.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Percent (%) Change in Levels of pS6, pAKt473, and Ki-67
Time Frame: 21 days post treatment with rapamycin
Population: paraffin embedded formalin fixed tissues including head and neck cancer lesion were not available for 2 participants
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Sirolimus
Number analyzed (Participants) | 14
percentage of change from baseline
  pS6 | -60.60 (18.71)
  pAKt473 | -67.24 (34.28)
  Ki-67 | -31.48 (35.47)
  pERK | 100.00 (104.95)

2. Primary Outcome: Percent (%) Changes in Tumor Size, Blood Flow, and Standardized Uptake Value
Time Frame: 21 days post treatment with rapamycin
Population: It was not possible to obtain appropriate CT scans or SUV measurement from all participants
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Sirolimus
Number analyzed (Participants) | 14
percentage change from baseline
  Tumor size by CT | -15.75 (26.46)
  SUV non-nodal target lesions: number analyzed (Participants) | 12
  SUV non-nodal target lesions | -31.84 (27.90)
  SUV lymph nodes: number analyzed (Participants) | 11
  SUV lymph nodes | -48.01 (23.67)

3. Primary Outcome: Percent (%) Change in Clinical and Laboratory Evaluations for Safety
Time Frame: Percent (%) change from Pre to Post treatement (~21 days)
Population: Same sample loss during processing for phosphor and magnesium
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
percentage change from baseline
  ANC | -45.51 (13.456)
  HCT | -5.71 (6.141)
  HGB | -5.32 (6.747)
  MCH | -2.53 (1.328)
  MCHC | 0.38 (2.090)
  MCV | -2.88 (1.399)
  MPV | -0.85 (5.149)
  PLAT | -25.10 (18.045)
  RBC | -2.87 (6.920)
  RDW | -5.19 (2.909)
  WBC | -32.31 (11.911)
  BUN | -0.00 (32.782)
  Ca | -4.80 (2.329)
  Cl | -0.25 (2.925)
  CO2 | -1.26 (8.261)
  CREATININE | -3.31 (10.397)
  GLUCOSE | 16.28 (37.433)
  K | -3.55 (9.259)
  Mg: number analyzed (Participants) | 15
  Mg | -4.22 (7.691)
  Na | -0.60 (1.933)
  PHOSPHOR: number analyzed (Participants) | 14
  PHOSPHOR | -6.58 (16.324)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of consent to one year post treatment.
Description: Subjects were followed 360 days after treatment, surgical or chemo radiation, to assess survival, recurrence of disease, metastases and adverse events that were related to rapamycin therapy including complications of wound healing, infections due to immune compromise and late radiation toxicities.
Arm/Group | Sirolimus
Serious Adverse Events (participants affected / at risk) | 3/16
Other Adverse Events (participants affected / at risk) | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus (N=16)
Injury, procedural complications/post-operative wound complication (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Subject had an active bleed from the original tonsillectomy site intraoperative which necessitated extended intubation to postoperative Day 2 when the subject was successfully extubated without further bleeding or complications.
Injury, procedural complications/postoperative wound complication (Infections and infestations) | 1 (2) — Orocutaneous fistula with left leg epidermolysis. Jaw hardware candida infection, surgical flap necrosis/failure.
Cardiac Disorder (Cardiac disorders) | 1 (1) — Left Bundle Branch Block diagnosed on routine stress test. Subject had left heart catheterization with stent placement.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus (N=16)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (8) — Thrombocytopenia Neutropenia Anemia Leukopenia
Investigations (Investigations) | 7 (7) — Combined decreased: neutrophil count, phosphorous, potassium, white blood cell, platelet. Combined increased: ALT, AST. BUN, glucose, BUN, hepatic enzymes, monocyte count
Gastrointestinal disorders (Gastrointestinal disorders) | 3 (3) — Combined events reported: vomiting, dysphagia, nausea, oral pain
Nervous system disorders (Nervous system disorders) | 3 (3) — Combined headache, dizziness, hypogeusia
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Combined: oropharyngeal pain, nasal congestion
General Disorders and administration site conditions (General disorders) | 2 (2) — Combined: mucosal inflammation, pain, pyrexia
Injury, poisoning, and procedural complications (Injury, poisoning and procedural complications) | 2 (2) — Combined: postoperative wound complications and post procedural hemorrhage
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 (2) — Combined: dehydration, hyperglycemia, hypoalbuminaemia
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 (2) — Combined: photosensitivity and rash
Cardiac disorders (Cardiac disorders) | 1 (1) — Coronary artery disease

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes